CLINICAL TRIAL: NCT03012204
Title: Series Study About the rTMS Effects on the Recovery of Limb Motor Dysfunction Due to Cerebral Vascular Disease, Part 1: Comparing the Effects of Various Combinations Between 6 Hertz(Hz) rTMS & LFrTMS.
Brief Title: Comparing Effects of Various Combinations of 6 Hertz(Hz) rTMS & LFrTMS on Motor Recovery Due to Cerebrovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, ZHUANG Li, MD, Chief Physician, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-2016010
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Cerebrovascular Disease
Keywords: Cerebrovascular Disease; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- combined rTMS at both M1 (Experimental): combined rTMS at both M1: sham 6 hertz(Hz) rTMS on unaffected M1 / real 1 Hz rTMS on unaffected M1 / real 6 Hz rTMS on affected M1
  Interventions: Device: combined rTMS at both M1
- real primed LFrTMS at unaffected M1 (Experimental): real primed LFrTMS at unaffected M1: real 6 hertz(Hz) rTMS on unaffected M1 / real 1 Hz rTMS on unaffected M1 / sham 6 Hz rTMS on affected M1
  Interventions: Device: real primed LFrTMS at unaffected M1
- real LFrTMS at unaffected M1 (Active Comparator): real LFrTMS at unaffected M1: sham 6 hertz(Hz) rTMS on unaffected M1 / real 1 Hz rTMS on unaffected M1 / sham 6 Hz rTMS on affected M1
  Interventions: Device: real LFrTMS at unaffected M1
- all sham stimulation (Sham Comparator): all sham stimulation： sham 6 hertz(Hz) rTMS on unaffected M1 / sham 1 Hz rTMS on unaffected M1 /sham 6 Hz rTMS on affected M1
  Interventions: Device: all sham stimulation

INTERVENTIONS:
Device: real LFrTMS at unaffected M1 — Compare the effect of LFrTMS at unaffected M1 to that of all sham stimulation on motor rehabilitation after cerebrovascular disease .
  rTMS: Repetitive Transcranial Magnetic Stimulation. Combination Elements: ①6 hertz(Hz) rTMS at unaffected M1 before LFrTMS at unaffected M1 ;②6 Hz rTMS at affected M1;③1 Hz rTMS at unaffected M1.
  The four groups are the combinations of real or sham ①/②/③.
  Arms: real LFrTMS at unaffected M1
Device: real primed LFrTMS at unaffected M1 — Compare the effect of primed LFrTMS at unaffected M1 to that of LFrTMS at unaffected M1 on motor rehabilitation after cerebrovascular disease .
  rTMS: Repetitive Transcranial Magnetic Stimulation. Combination Elements: ①6 hertz(Hz) rTMS at unaffected M1 before LFrTMS at unaffected M1 ;②6 Hz rTMS at affected M1;③1 Hz rTMS at unaffected M1.
  The four groups are the combinations of real or sham ①/②/③.
  Arms: real primed LFrTMS at unaffected M1
Device: combined rTMS at both M1 — Compare the effect of combined rTMS at both M1 to that of primed LFrTMS at unaffected M1 on motor rehabilitation after cerebrovascular disease .
  rTMS: Repetitive Transcranial Magnetic Stimulation. Combination Elements: ①6 hertz(Hz) rTMS at unaffected M1 before LFrTMS at unaffected M1 ;②6 Hz rTMS at affected M1;③1 Hz rTMS at unaffected M1.
  The four groups are the combinations of real or sham ①/②/③.
  Arms: combined rTMS at both M1
Device: all sham stimulation — used as controls to eliminate the placebo effect of all kinds of combinated rTMS
  Arms: all sham stimulation

SUMMARY:
To compare the effects of various combinations between 6 hertz(Hz) rTMS & LFrTMS on the limb motor dysfunction due to cerebral vascular disease.

DETAILED DESCRIPTION:
It is the basic principle for functional recovery after cerebrovascular disease to restore the original balance in reciprocal inhibition between affected hemisphere and unaffected hemisphere.

repetitive transcranial magnetic stimulation (rTMS) is a noninvasive neuroplastic technique rebalancing interhemispheric competition after stroke. Low frequency rTMS (LFrTMS) on contralesional hemisphere or high frequency rTMS (HFrTMS) on lesional hemisphere might be the basic choice.

6 hertz(Hz) primed LFrTMS on lesional primary motor cortex has the stronger effect than LFrTMS alone does on one hand; the other newly-developed combination, i.e. HFrTMS on lesional primary motor cortex and LFrTMS on contralesional primary motor cortex might also be more effective than they do respectively on the other hand.

The main aim of our research is to find out which combination is better by considering both safety and efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 30 to 90 years;
* Newly onset cerebral infarction or brain hemorrhage confirmed by MRI or CT;
* the disease duration is less than 20 weeks when recruited into the trial;
* no existence of limb motor dysfunction before this onset, and new occurrence of unilateral limb motor dysfunction after this onset;
* the physical and mental condition are good enough to cooperate with the assessment and treatment;
* the NIHSS score: total 5-20,1a,1b,1c=0;
* the subject or legal guardian sign the consent form.

Exclusion Criteria:

* during pregnancy;
* with skull defect;
* with metal implants, cardiac pacemaker, cochlear implantation;
* epileptiform discharge in EEG.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer assessment (FMA) | 1) Before treatment (Baseline); 2) Change from Baseline FMA at the 1st workday after the last treatment; 3) Change from Baseline FMA at the 28th natural day after the last treatment
  Score of Fugl-Meyer assessment
Simple Test for Evaluating Hand Function (STEF) | 1) Before treatment (Baseline); 2) Change from Baseline STEF at the 1st workday after the last treatment; 3) Change from Baseline STEF at the 28th natural day after the last treatment
  Score of Simple Test for Evaluating Hand Function

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | 1) Before treatment (Baseline); 2) Change from Baseline NIHSS at the 1st workday after the last treatment; 3) Change from Baseline NIHSS at the 28th natural day after the last treatment
  Score of National Institute of Health Stroke Scale

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhuang, M.D., Principal Investigator — Beijing Hospital, National Center of Gerontology, China
Locations (1):
- Beijing Hospital, National Center of Gerontology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sung WH, Wang CP, Chou CL, Chen YC, Chang YC, Tsai PY. Efficacy of coupling inhibitory and facilitatory repetitive transcranial magnetic stimulation to enhance motor recovery in hemiplegic stroke patients. Stroke. 2013 May;44(5):1375-82. doi: 10.1161/STROKEAHA.111.000522. Epub 2013 Mar 26. PMID 23532011
- [Background] Wang CP, Tsai PY, Yang TF, Yang KY, Wang CC. Differential effect of conditioning sequences in coupling inhibitory/facilitatory repetitive transcranial magnetic stimulation for poststroke motor recovery. CNS Neurosci Ther. 2014 Apr;20(4):355-63. doi: 10.1111/cns.12221. Epub 2014 Jan 15. PMID 24422912
- [Background] Carey JR, Anderson DC, Gillick BT, Whitford M, Pascual-Leone A. 6-Hz primed low-frequency rTMS to contralesional M1 in two cases with middle cerebral artery stroke. Neurosci Lett. 2010 Jan 29;469(3):338-42. doi: 10.1016/j.neulet.2009.12.023. Epub 2009 Dec 18. PMID 20026185
- [Background] Cassidy JM, Chu H, Anderson DC, Krach LE, Snow L, Kimberley TJ, Carey JR. A Comparison of Primed Low-frequency Repetitive Transcranial Magnetic Stimulation Treatments in Chronic Stroke. Brain Stimul. 2015 Nov-Dec;8(6):1074-84. doi: 10.1016/j.brs.2015.06.007. Epub 2015 Jun 22. PMID 26198365
- [Background] Carey JR, Evans CD, Anderson DC, Bhatt E, Nagpal A, Kimberley TJ, Pascual-Leone A. Safety of 6-Hz primed low-frequency rTMS in stroke. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):185-92. doi: 10.1177/1545968307305458. Epub 2007 Sep 17. PMID 17876070